CLINICAL TRIAL: NCT03865472
Title: Enhancing Relapse Prevention With rTMS: Dose-Response Parameters for Smoking Cessation
Brief Title: rTMS in Promoting Smoking Cessation and Preventing Relapse in Current Smokers
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Roswell Park Cancer Institute (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: i 65718; NCI-2018-03300 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); i 65718 (Other: Roswell Park Cancer Institute); R01CA229415 (NIH)
Record Dates: First submitted 2019-03-04; First posted 2019-03-07 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Cigarette Smoker; Current Every Day Smoker; Current Smoker
MeSH Terms: interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm I (rTMS) (Experimental): Patients undergo rTMS QD or BID over 16 minutes for 8, 12, or 16 days.
  Interventions: Other: Questionnaire Administration; Procedure: Repetitive Transcranial Magnetic Stimulation
- Arm II (sham rTMS) (Sham Comparator): Patients undergo sham rTMS QD or BID over 16 minutes for 8, 12, or 16 days.
  Interventions: Other: Questionnaire Administration; Procedure: Sham Intervention

INTERVENTIONS:
Other: Questionnaire Administration — Ancillary studies
Procedure: Repetitive Transcranial Magnetic Stimulation — Undergo rTMS
  Other Names: rTMS
  Arms: Arm I (rTMS)
Procedure: Sham Intervention — Undergo sham rTMS
  Arms: Arm II (sham rTMS)

SUMMARY:
This trial studies best dose and how well repetitive transcranial magnetic stimulation (rTMS) works in promoting smoking cessation and preventing relapse in current smokers. rTMS is a form of brain stimulation therapy that controls nerve cell activity, increases blood flow in the brain, and improves cognitive function.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To examine the effects of stimulation duration (stimulation days) and intensity (pulses per day) on outcomes among smokers (sample size [n]=258) motivated to quit.

II. To identify the most promising dosing strategy by balancing effect sizes and undesirable effects.

III. To examine the effects of 16 20Hz rTMS sessions combined with intensive cognitive behavioral treatment and nicotine replacement on smoking cessation, developmental disability (DD rates), cognitive behavioral skill acquisition, and nicotine patch adherence among lung cancer (LC) patients (n=30). (Study 1 and Study 2) IV. To examine the feasibility and potential efficacy of 20Hz rTMS on the left dorsolateral prefrontal cortex (DLPFC) for concurrent smoking abstinence and reductions in alcohol use among smokers who are heavy drinkers (n=20). (Study 1 and Study 2)

OUTLINE: Patients are randomized to 1 of 2 arms.

ARM I: Patients undergo rTMS once daily (QD) or twice daily (BID) over 16 minutes for 8, 12, or 16 days.

ARM II: Patients undergo sham rTMS QD or BID over 16 minutes for 8, 12, or 16 days.

ELIGIBILITY:
Inclusion Criteria:

* Participants will be right-handed
* Negative urine drug screen at the baseline assessment
* Ability to read at the 8th grade level
* Passes the Transcranial Magnetic Stimulation Adult Safety and Screening Questionnaire (TASS)
* Participants must smoke between 5 and 25 cigarettes per day with the intent to quit smoking in the next 30 days
* Participant or legal representative must understand the investigational nature of this study and sign an Independent Ethics Committee/Institutional Review Board approved written informed consent form prior to receiving any study related procedure
* Study 1: Participants will be right-handed and have been diagnosed with primary non-small and small cell lung cancer or with non-skin squamous cell HNC (self-reported)
* Study 1: Age 18+
* Study 1: Negative urine drug screen at the baseline assessment
* Study 1: Ability to read at the 8th grade level
* Study 1: Passes the Transcranial Magnetic Stimulation Adult Safety and Screening Questionnaire (TASS)
* Study 1: Participants must smoke at least 4 cigarettes per day and intend to quit smoking in the next 60 days
* Study 1: Has been diagnosed with primary non-small cell LC or with primary non-skin squamous cell HNC (self-reported)
* Study 2: Participants will be healthy right-handed adults
* Study 2: Age 18-65 years old
* Study 2: Negative urine drug screen at the baseline assessment
* Study 2: Ability to read at the 8th grade level
* Study 2: Passes the Transcranial Magnetic Stimulation Adult Safety and Screening Questionnaire (TASS)
* Study 2: Participants must smoke between 5 and 25 cigarettes per day with the intent to quit smoking in the next 30 days
* Study 2: Meet the criteria for heavy alcohol use: > 7 drinks per week for women, > 15 drinks per week for men OR binge drinking >= 5 days in the past month. Binge drinking is defined as >= 4 drinks for women and >= 5 drinks for men, consumed within 2 hours of each other
* Study 2: Participant or legal representative must understand the investigational nature of this study and sign an Independent Ethics Committee/Institutional Review Board approved written informed consent form prior to receiving any study related procedure

Exclusion Criteria:

* Has a personal history of epilepsy
* Has a history of anticonvulsant medication use
* Has a personal history of head injury
* Has a History of aneurysm, stroke, or previous cranial neurosurgery or abnormal findings on the magnetic resonance imaging (MRI) (e.g., tumor, aneurism, etc.)
* Has uncontrolled major depressive disorder, bipolar disorder or a schizophrenia-spectrum disorder, or tinnitus
* Has any metal implants or neuro-stimulators in the head, neck, or cochlea that prevent an MRI being performed
* Has a pacemaker
* Personal history of migraine headaches
* Currently taking medications that lower seizure threshold (e.g., such as tricyclic antidepressants or bupropion)
* Currently using medications for tobacco cessation (e.g., nicotine replacement, bupropion, varenicline, etc)
* Pregnant or planning to become pregnant in the next 24 weeks
* Current regular use of forms of tobacco other than cigarettes including e-cigarettes
* Participants who score above 48.3 on the Claustrophobia Questionnaire at the baseline assessment will be excluded because they are likely to be unable to undergo an magnetic resonance imaging (MRI) without distress
* Individuals who score >15, indicative of moderate-severe Alcohol Use Disorder, on the Alcohol Use Disorders Identification Test (AUDIT).
* Unwilling or unable to follow protocol requirements
* Any condition which in the Investigator's opinion deems the participant an unsuitable candidate to participate in the study

  * Study 1:Has a personal history of Brain metastases
  * Study 1: Unable to use nicotine patches
  * Study 1: Has a Personal history of epilepsy
  * Study 1: Has a History of anticonvulsant medication use
  * Study 1: Has a Personal history of head injury
  * Study 1: History of aneurysm, stroke, or previous cranial neurosurgery or abnormal findings on the MRI (e.g., tumor, aneurism, etc.)
  * Study 1: A diagnosis of major depressive disorder, bipolar disorder or a schizophrenia-spectrum disorder, or tinnitus
  * Study 1: Has any Metal implants or neuro-stimulators in the head, neck, or cochlea that prevent an MRI being performed
  * Study 1: Has a pacemaker
  * Study 1: Personal history of Migraine headaches
  * Study 1: Currently taking medications that lower seizure threshold (e.g., such as tricyclic antidepressants or bupropion)
  * Study 1: Currently using bupropion or varenicline for smoking cessation
  * Study 1: Pregnant or planning to become pregnant in the next 24 weeks
  * Study 1: Current regular use of forms of tobacco other than cigarettes
  * Study 1: Participants who score above 48.3 on the Claustrophobia Questionnaire at the baseline assessment will be excluded because they are likely to be unable to undergo a magnetic resonance imaging (MRI) scan without distress
  * Study 1: Unwilling or unable to follow protocol requirements
  * Study 1: Any condition which in the Investigator's opinion deems the participant an unsuitable candidate to participate in the study
  * Study 2: Has a personal history of epilepsy
  * Study 2: Has a history of anticonvulsant medication use
  * Study 2: Has a personal history of head injury
  * Study 2: Has a history of aneurysm, stroke, or previous cranial neurosurgery or abnormal findings on the MRI (e.g., tumor, aneurism, etc.)
  * Study 2: Has a diagnosis of major depressive disorder, bipolar disorder or a schizophrenia-spectrum disorder, or tinnitus
  * Study 2: Has any metal implants or neuro-stimulators in the head, neck, or cochlea that prevent an MRI being performed
  * Study 2: Has a pacemaker
  * Study 2: Personal history of Migraine headaches
  * Study 2: Currently taking medications that lower seizure threshold (e.g., such as tricyclic antidepressants or bupropion)
  * Study 2: Currently using medications for tobacco cessation (e.g., nicotine replacement, bupropion, varenicline, etc.)
  * Study 2: Pregnant or planning to become pregnant in the next 24 weeks
  * Study 2: Current regular use of forms of tobacco other than cigarettes
  * Study 2: Participants who score above 48.3 on the Claustrophobia Questionnaire at the baseline assessment will be excluded because they are likely to be unable to undergo a magnetic resonance imaging (MRI) without distress
  * Study 2: Meet the criteria for severe alcohol use disorder (AUD) (> 6 symptoms) or have ever met Diagnostic and Statistical Manual of Mental Disorders-Fifth Edition (DSM-V) criteria for alcohol withdrawal. Heavy drinking and AUD are not mutually exclusive.
  * Study 2: Unwilling or unable to follow protocol requirements
  * Study 2: Any condition which in the Investigator's opinion deems the participant an unsuitable candidate to participate in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 206 (Actual)
Dates: Start 2018-11-10 (Actual); Primary Completion 2025-11-13 (Actual); Study Completion 2026-11-13 (Estimated)

PRIMARY OUTCOMES:
Latency to relapse | Up to 30 days
  Latency to relapse will be defined as the number of days from the quit day to relapse. Relapse will be defined as smoking for seven consecutive days. Will use Cox proportional-hazards (CPH) models to examine latency to relapse outcome. Ties in failure times will be handled using methods developed by Efron. Compliance with the CPH assumptions will be tested by coding the factors as time-dependent covariates.

SECONDARY OUTCOMES:
Point-prevalence abstinence rates | At 12 and 24 weeks after quit date
  Will use logistic regression models to examine binary 12 and 24-week point prevalence abstinence.
Delay discounting rates | At 12 and 24 weeks after quit date
  Will be examined through using repeated measures Generalized Linear models.
Cognitive-behavioral Therapy Skills Questionnaire | Up to 24 weeks
  Cognitive behavioral skills will be assessed using the Cognitive-Behavioral Therapy Skills Questionnaire (CBTSQ)
Side effects | Up to 24 weeks
  Potential undesirable effects will be measured up to 24 weeks.
Forever Free (FF) Booklet content Exposure | Up to 24 weeks
  Will be measured in terms of number of content segments in each booklet.

CONTACTS AND LOCATIONS:
Overall Officials: Christine Sheffer, Principal Investigator — Roswell Park Cancer Institute
Locations (1):
- Roswell Park Cancer Institute, Buffalo, New York, United States

REFERENCES:
- [Derived] Shevorykin A, Carl E, Liskiewicz A, Hanlon CA, Bickel WK, Mahoney MC, Vantucci D, Bensch L, Thorner H, Marion M, Sheffer CE. Perceived research burden of a novel therapeutic intervention: A study of transcranial magnetic stimulation for smoking cessation. Front Rehabil Sci. 2023 Mar 3;4:1054456. doi: 10.3389/fresc.2023.1054456. eCollection 2023. PMID 36937103
- [Derived] Shevorykin A, Carl E, Mahoney MC, Hanlon CA, Liskiewicz A, Rivard C, Alberico R, Belal A, Bensch L, Vantucci D, Thorner H, Marion M, Bickel WK, Sheffer CE. Transcranial Magnetic Stimulation for Long-Term Smoking Cessation: Preliminary Examination of Delay Discounting as a Therapeutic Target and the Effects of Intensity and Duration. Front Hum Neurosci. 2022 Jul 5;16:920383. doi: 10.3389/fnhum.2022.920383. eCollection 2022. PMID 35874156
- [Derived] Carl E, Liskiewicz A, Rivard C, Alberico R, Belal A, Mahoney MC, Quisenberry AJ, Bickel WK, Sheffer CE. Dosing parameters for the effects of high-frequency transcranial magnetic stimulation on smoking cessation: study protocol for a randomized factorial sham-controlled clinical trial. BMC Psychol. 2020 May 1;8(1):42. doi: 10.1186/s40359-020-00403-7. PMID 32357940

DOCUMENTS (1):
  • Informed Consent Form (2025-04-15): https://cdn.clinicaltrials.gov/large-docs/72/NCT03865472/ICF_000.pdf